CLINICAL TRIAL: NCT05198752
Title: A Phase 1 Clinical Study to Evaluate the Tolerability, Safety,Immunogenicity and Efficacy of the Neoantigen mRNA Personalised Cancer Vaccine SW1115C3 in Patients With Advanced Malignant Solid Tumours
Brief Title: A Study of Neoantigen mRNA Personalised Cancer in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stemirna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SWP1001-06
Record Dates: First submitted 2022-01-05; First posted 2022-01-20 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Solid Tumor

STUDY DESIGN:
Intervention Model Description: 30 participants in Cohort (C)1:50 mcg of SW1115C3 ; C2: 100 mcg of SW1115C3; C3: 150 mcg of SW1115C3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoantigen mRNA Personalised Cancer (Experimental): This study is a 3+3 dose escalation design. Participants will receive a total of 6 cycles of SW1115C3 every 21 days.
  Interventions: Drug: Neoantigen mRNA Personalised Cancer SW1115C3

INTERVENTIONS:
Drug: Neoantigen mRNA Personalised Cancer SW1115C3 — Subcutaneous Injection

SUMMARY:
This is a Phase 1 open label study to evaluate the tolerability, safety, immunogenicity, and efficacy of SW1115C3, a neoantigen mRNA personalised cancer vaccine, in patients with advanced malignant solid tumours.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 to 80 years old (including boundary values), without limitation of sex at time of consent.
* Based on the RECIST 1.1 criteria for disease progression, (a maximum increase in tumour diameter of 20%) for participants undergoing prescreening who are receiving standard treatment, these participants may reach the defined disease progression criteria at the time of tumour vaccine administration.

Exclusion Criteria:

* Have used a live attenuated vaccine within 4 weeks before the first use of SW1115C3 with the following exceptions:
* Adverse reactions induced by previous anti-tumour treatments have not yet recovered to Grade ≤ 1 (except for toxicity evaluated to have no risk of safety by the PI [or designee], such as hair loss, Grade 2 peripheral neurotoxicity and hypothyroidism stabilised by hormone-replacement therapy) based on NCI CTCAE version 5.0.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2023-12-22 (Estimated); Study Completion 2024-06-12 (Estimated)

PRIMARY OUTCOMES:
，Dose-limiting toxicity incidence (participants who experience DLT) | 21 day

SECONDARY OUTCOMES:
Objective response rate(ORR) assessment per RECIST Version 1.1 | 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (2):
  - Pindara Private Hospital, Benowa, Queensland
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
- One Clinical Research, Nedlands, Western Australia, Austria

IPD SHARING:
Plan to Share IPD: No